CLINICAL TRIAL: NCT05094063
Title: The Effect of Education Supported by the Mobile Application Given to Patients Undergoing Open Heart Surgery on Postoperative Recovery and Psychological Well-Being of Patients
Brief Title: Patient Education by Mobile Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Betul Zeynep Yildiz (Other)
Responsible Party: Sponsor-Investigator, Betul Zeynep Yildiz, Principal Investigator, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/03-41
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Open Heart Surgery Patients
Keywords: open heart surgery; surgical nursing; patient education

STUDY DESIGN:
Intervention Model Description: This research was planned as an experimental randomized controlled trial. Randomization will be done using a computer program. With the computer program (www.randomizer.org), the participants will be divided into 2 subgroups (group 1: patient education group; group 2: patient education group not provided). With the randomization program, the order of the experimental and control groups will be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Training will be given to the patients in the experimental group.
  Interventions: Other: patient education by mobile application
- control group (No Intervention): untrained patient group

INTERVENTIONS:
Other: patient education by mobile application — Training will be given to the patients in the experimental group.
  Arms: experimental group

SUMMARY:
Cardiovascular diseases are among the important health problems that cause mortality and morbidity both in our country and in the World (Sidar vd 2013). According to the data of the Turkish Statistical Institute (2021), circulatory system diseases were the first cause of mortality in our country in 2018 with a rate of 38.4%. According to the data of the World Health Organization, the disease that causes the most death in the world is ischemic heart disease with 16% (World Health Organization,2021).

In addition to acute care, the aim of education in patients with cardiovascular surgery is to support patients' self-care and post-operative recovery, to enable patients and their families to self-manage their care at home, to reduce postoperative complications and rehospitalization rates(Akyolcu vd 2017).

Training can be delivered using a combination of formats including brochures, online, books, audio cassette, videotape, and/or skype (Fredericks & Yau, 2012). Booklets, brochures, tele-health, and web design methods were used in the training given to patients who had heart surgeries in previous years in our country.

In this study, the training booklet to be used in the education to be given to the patients will be prepared by the researchers. The content of the prepared training booklet will be presented to patients in the form of a mobile application that can run on smart phones with Android operating system so that patients can follow it. With this research, it is aimed to facilitate access to information and accelerate post-operative recovery. In the future, this practice will also contribute to reducing stationery costs.

DETAILED DESCRIPTION:
In this study, the training booklet to be used in the education to be given to the participants will be prepared by the researchers. In addition, the content of the prepared training booklet will be presented to participants in the form of a mobile application that can run on smart phones with Android operating system so that participants can follow it. In the content of the mobile application, there will be an interface with the information in the booklet and the video narration of the exercises that the participants should do. This application will be downloadable through the server and then there will be no internet requirement to use the application. The mobile application will be installed on the participants' own phones. The participants will be able to adjust the font size in the application. The participants will see the titles in the booklet and will reach the information by choosing the subject curious about. Participants will also be able to listen to the information in the booklet in the form of an audio recording. In addition, reminder notifications for medications and exercises will be set for participants in the mobile application. In this way, it will be easier for participants to access information, and it will be ensured that participants do not forget participants medication hours and that they do the exercises participants need to do during the day without forgetting. Every day between 18.30-20.30, a questionnaire will be sent to the user to evaluate the amount/time of exercise participants has applied for that day. Thus, it will be ensured that the answers of the participants are sent to the server and the daily follow-up of the participants will be carried out. The device will need internet access to send information. The information sent will be kept on the database and can be easily processed. However, it will be possible to easily access the user's historical information without data confusion. It is planned to store the data on MySql (My Structured Query Language) database. If any update is required to the application, it will be carried out quickly through the server. After the research, the use of the mobile application will be continued and sustainability will be ensured in the postoperative recovery and psychological well-being of the participants.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily accepting to participate in the study
* 18 years and over
* Having planned surgery
* Conscious Open
* Coming to the clinic from the intensive care unit after the operation
* Having no vision, hearing and speech problems
* Stable clinical condition
* Able to communicate
* Having a phone with Android operating system (for the experimental group)
* Patients without a psychiatric history

Exclusion Criteria:

* Cancellation of the operation
* Inability to communicate with the patient
* The patient's desire to withdraw from the study
* Deterioration of the patient's clinical condition
* The patient's inability to use the mobile application

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Postoperative Recovery Index (PoRI) at month 3 | Baseline and month 3
  There are 5 sub-dimensions of PoRI; psychological symptoms, physical activities, general symptoms, intestinal symptoms, and craving-desire symptoms. The scores of the items included in the sub-dimensions are summed, their arithmetic average is taken, and the sub-dimension score is determined. A minimum of 1 and a maximum of 5 points can be obtained from the PoRI. High scores from the index reflect more difficulty in post-operative recovery, while low scores indicate that post-operative recovery is easier.
Change from baseline in Psychological Well-Being at month 3 | Baseline and month 3
  Flourishing Scale (FS), which is a psychological well-being scale in Turkish identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life. The items of FS are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). A minimum of 8 and a maximum of 56 points can be obtained from the FS. A high score indicates that the person has many psychological resources and strengths.

SECONDARY OUTCOMES:
Change from baseline in StateTrait Anxiety Inventory at month 3 | Baseline and month 3
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Fredericks S, Yau TM. Educational interventions for adults to prevent readmission and complications following cardiovascular surgery. Cochrane Database of Systematic Reviews 2012, Issue 9.
- [Background] Sidar A , Dedeli Ö, İşkesen Aİ. The Relationship Between Anxiety, Pain Distress and Pain Severity Before and After Open Heart Surgery in Patients Yoğun Bakım Derg, 2013, 4: 1-8.
- [Background] Akyolcu N, Kanan N, Güler A. Cerrahi Hemşireliği II, 1. Baskı. İstanbul, Nobel Tıp Kitapevleri, 2017: 101-114.
- See also: WHO internet web site — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death